CLINICAL TRIAL: NCT06290115
Title: Relationship Between Non-suicidal Self-injury Behaviors in Adolescents and Young Adults and Perceived Parental Negative Emotional Expression and Family Communication Styles in Children:A Case-control Study
Brief Title: Adolescents' Non-suicidal Behavior and Perception of Parents' Negative Emotional Expression and Family Communication
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, associate professor, Sun Yat-sen University
Other Study IDs: 202301
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Adolescents
Keywords: Adolescents and Young Adults; Non-suicidal self-injury; Parental emotional expressivity; Family communication patterns
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case group: NSSI patient group: 1. Patients who meet the diagnostic criteria in DSM-5 and are clinically diagnosed as NSSI;
  2. Age range: 15-25 years old;
  3. Clear consciousness, normal speech function, able to communicate in Chinese and reading chinese;
  Interventions: Other: Questionnaires set 1
- Control group 1: non-NSSI patients: 1. psychiatric outpatients or inpatients can read and understand the contents of the questionnaire;
  2. Patients who do not meet the diagnostic criteria in DSM-5 and are clinically diagnosed as NSSI.
  3. Age range: 15-25 years old;
  4. Clear consciousness, normal speech function, able to communicate in Chinese and reading chinese;
  Interventions: Other: Questionnaires set 2
- Control group 2: healthy group: 1. No mental illness;
  2. Age range: 15-25 years old;
  3. Clear consciousness, normal speech function, able to communicate in Chinese and reading chinese;
  Interventions: Other: Questionnaires set 3

INTERVENTIONS:
Other: Questionnaires set 1 — Participants of case group will be asked to respond to the demographic information，the Family Emotional Expressivity Questionnaire（FEEQ）、the Parent-Adolescent Communication Scale（PACS）、the Childhood Trauma Questionnaire（CTQ）、the Parental Bongding Instrument（PBI）、the Adolescent parent-child relationship intimacy questionnaire and the Ottawa Self-injury Inventory（OSI）.
  Groups: Case group: NSSI patient group
Other: Questionnaires set 2 — Participants of control group 1 will be asked to respond to the demographic information，the Family Emotional Expressivity Questionnaire（FEEQ）、the Parent-Adolescent Communication Scale（PACS）、the Childhood Trauma Questionnaire（CTQ）、the Parental Bongding Instrument（PBI） and the Adolescent parent-child relationship intimacy questionnaire.
  Groups: Control group 1: non-NSSI patients
Other: Questionnaires set 3 — Participants of control group 2 will be asked to respond to the demographic information，the Family Emotional Expressivity Questionnaire（FEEQ）、the Parent-Adolescent Communication Scale（PACS）、the Childhood Trauma Questionnaire（CTQ）、the Parental Bongding Instrument（PBI） and the Adolescent parent-child relationship intimacy questionnaire.
  Groups: Control group 2: healthy group

SUMMARY:
The starting point of this project is to study young people and adolescents, aiming to explore the correlation between non-suicidal behavior of young people and adolescents and the negative emotional expression of their parents and family communication. The purpose of this project is to investigate the non-suicidal self-injury behavior of teenagers aged 15-25 years by issuing questionnaires (sample size: 327 people). In order to find out whether there is any connection between family communication and non-suicidal self-injury behavior of young people and adolescents.

DETAILED DESCRIPTION:
The incidence of non-suicidal self-injury（NSSI） among adolescents has obviously increased, which should attract the attention of the whole society. Their mental health problems will not only lead to personal pain and family burden, but also bring potential negative effects to future social development. Therefore, it is necessary to study the psychological problems of teenagers and their influencing factors. This study will conduct a case-control study from the perspective of family, and analyze the negative emotional expression and family communication style of parents of non-suicidal teenagers and their influence on non-suicidal self-injury behavior. This study is conducted in the form of scale, which will use the demographic information，the Family Emotional Expressivity Questionnaire（FEEQ）、the Parent-Adolescent Communication Scale（PACS）、the Childhood Trauma Questionnaire（CTQ）、the Parental Bongding Instrument（PBI）、the Adolescent parent-child relationship intimacy questionnaire and the Ottawa Self-injury Inventory（OSI）.

ELIGIBILITY:
1.Case group: NSSI patient group:

Inclusion Criteria:

1. Patients who meet the diagnostic criteria in DSM-5 and are clinically diagnosed as NSSI;
2. Age range: 15-25 years old;
3. Clear consciousness, normal speech function, able to communicate in Chinese and reading chinese;

Exclusion Criteria:

1. Users with organic diseases and psychoactive substances;
2. NSSI； caused by autism, TIC disorder, mental retardation and other emotional instability and bad mood;
3. Religious self-injury or customary self-injury;
4. Patients with schizophrenia, schizoaffective disorder, alcohol dependence, organic mental disorder and other mental disorders have been previously diagnosed.

2.Control group 1: Non-NSSI patients

Inclusion criteria:

1. Psychiatric outpatients or inpatients can read and understand the contents of the questionnaire;
2. Patients who do not meet the diagnostic criteria in DSM-5 and are clinically diagnosed as NSSI.
3. Age range: 15-25 years old;
4. Patients and/or guardians can give informed consent and participate in this study.

Exclusion criteria:

1. Patients whose illness causes them unable to communicate or fill out questionnaires;
2. Non-serious mental diseases, such as schizophrenia and schizoaffective disorder.

3.Control group 2: Healthy group

Inclusion criteria

1. No mental illness;
2. Age range: 15-25 years old;
3. Clear consciousness, normal speech function, able to communicate in Chinese and reading chinese;
4. Patients and/or guardians can give informed consent and participate in this study.

Exclusion criteria

(1) Young people and adolescents who are unable to communicate or fill out questionnaires due to various organic reasons.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The group of adolescents and young adults diagnosed as NSSI, and the control group includes adolescents and young adults with other mental diseases other than NSSI, healthy adolescents and young adults.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-suicidal self-injury behavior of young people and adolescents | Baseline
  There are 28 items in the Ottawa Self-injury Inventory, which are used to evaluate the frequency of NSSI and suicide in the last 1, 6 and 12 months, the age of first onset, the source and concealment of self-injury ideas, and the feeling of self-injury impulse.
Expression of negative emotions of parents | Baseline
  There are 40 items in the Parental Emotional Expression Questionnaire, which is used to measure parents' negative emotions. The scale adopts system, and the higher the dimension score, the greater the possibility of negative emotions.
Parent-Adolescent communication scale | Baseline
  There are 40 items in the parent-Adolescent communication scale, which is used to measure parent-child communication. The scale adopts Likert 5-point system, and the higher the score, the better the parent-child communication.

SECONDARY OUTCOMES:
Childhood Trauma Questionnaire | Baseline
  There are 28 items in the Childhood Trauma Scale, which are used to measure childhood traumatic experiences. The scale adopts Likert 5-point system, and the higher the score, the more serious the childhood trauma experience.
Parental Bongding Instrument | Baseline
  There are 23 items in the Parenting Style Scale, which is used to measure the parenting style. The scale adopts Likert 4-point system, which consists of three factors: caring, encouraging autonomy and controlling.
The parent-child relationship intimacy scale | Baseline
  There are 29 items in the parent-child relationship intimacy scale, which are used to measure the parent-child relationship. The scale adopts Likert 5-point system, and the higher the score, the higher the intimacy of parent-child relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No